CLINICAL TRIAL: NCT02480790
Title: Venous Thromboembolic Complications in Patients With Ovarian Cancer Compared to Patients With Benign Ovarian Tumours
Brief Title: Venous Thromboembolic Complications in Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery (Other)
Responsible Party: Sponsor-Investigator, Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: OV-VTE
Record Dates: First submitted 2015-05-30; First posted 2015-06-25 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Venous Thromboembolism; Ovarian Neoplasms; Ovarian Cancer; Deep Vein Thrombosis; Lung Embolism
MeSH Terms: conditions — Venous Thromboembolism; Ovarian Neoplasms; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue and also healthy tissue for comparison are taken at surgery. Blood samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with malignant disease: Patients with ovarian, tubar or primary peritoneal cancer
- Patients with benign disease: Patients with suspected ovarian cancer where the final pathologic diagnosis is benign

SUMMARY:
Objectives of the study are: To estimate the incidence of venous thromboembolism (VTE) in a cohort of women with suspected ovarian cancer and evaluate changes in the coagulation system in case of benign or malignant disease. The impact of changes in the coagulation system on disease prognosis will be evaluated.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a common complication after surgery. Deep-vein thrombosis (DVT) and pulmonary embolism (PE) constitute VTE. PE is often a consequence of DVT and it is a feared complication and the most common preventable cause of hospital death. VTE can be asymptomatic and can be detected by a compression ultrasound scan (CUS) of the legs and a Computer Tomography (CT) of the lungs. It is wellknown that cancer patients are at higher risk of developing VTE, the risk is approximately seven times higher than in the background population. A Danish study showed a significantly higher risk of death when VTE was diagnosed at the same time as the cancer diagnosis with a 12 % one year survival compared to 36 % in cancer patients without a history of VTE.

Approximately 600 women in Denmark are diagnosed with ovarian cancer every year and it is the forth most common cause of cancer death among Danish women. Earlier studies have found that up to 31 % of ovarian cancer women develop VTE as a consequence of the disease and/or the treatment. Very few studies have examined the incidence of VTE before treatment.

Methods: A Pulmonary CT-angiography is included in the routinely performed Fluorodeoxyglucose Positron Emission Tomography - Computer Tomography (FDG PET-CT) to reveal pulmonary embolism at time of first referral. Compressive ultrasound scan including Doppler flow of the lower extremities is performed four times from first referral and during a one-year follow up period to detect clinical or subclinical deep vein thrombosis (DVT) before and after initiation of treatment.

Blood and tissue samples are taken, prepared and stored at -80 degrees in the Danish Cancer-Biobank for later analyzes of coagulation markers.

Immune histochemical techniques will be use to demonstrate tissue factor (TF) in tumor tissue.

The objectives of the study are:

1. In a prospective study at Aalborg University Hospital to estimate the incidence of clinical and subclinical venous thromboembolism (VTE) in patients with suspected ovarian cancer before and after initiation of treatment. The impact of VTE on survival will be evaluated.
2. In the same prospective cohort the correlation between markers of coagulation and fibrinolysis and subclinical VTE, tumour burden and overall survival will be evaluated.
3. Evaluate the correlation between immunohistochemical demonstrated tissue factor (TF) in tumour tissue and circulating TF in peripheral blood and the relation to VTE and tumour burden.

ELIGIBILITY:
Inclusion Criteria:

Women referred to the Department of Gynaecology and Obstetrics, Aalborg University Hospital on suspicion of ovarian cancer can be included if they present with a RMI ≥ 200.

Exclusion Criteria:

1. Previous cancer (within previous 3 years) or concomitant cancer of any origin.
2. Known immunological connective tissue disease.
3. Treatment with heparin, low molecular weight heparin (LMWH) or vitamin K antagonist at the time of inclusion.
4. Lack of informed consent.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women referred to the outpatient clinic with suspected ovarian cancer, where the initial examinations with ultrasound scan and measurement of ca-125 in blood reveal a Risk Malignancy Index (RMI) ≥ 200 indicating a high risk of ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolism due to ovarian cancer | one year
  Compressive ultrasound scan of lower extremities and pulmonary CT-angiography

SECONDARY OUTCOMES:
Changes in the coagulation system in case of ovarian cancer | one year
  Analysis of blood samples
Impact of changes in the coagulation system on disease prognosis in ovarian cancer | one year
  Evaluation of classic and novel coagulation markers and their relation to prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Ole Thorlacius-Ussing, MD, DMSc, Principal Investigator — Department of Gastrointestinal Surgery, Aalborg University Hospital
Locations (1):
- Department of Gynecology and Obstetrics, Aalborg University Hospital, Aalborg, Denmark